CLINICAL TRIAL: NCT04189198
Title: A Randomized Controlled Trial : Comparison of 4% Articaine Versus 0.5% Bupivacaine for Ambulatory Orthopaedic Surgery Under Supraclavicular Block
Brief Title: A Comparison of 4% Articaine Versus 0.5%Bupivacaine for Ambulatory Surgery Under Supraclavicular Block
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, simon Halim Armanious, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Articaine versus bupivacain
Record Dates: First submitted 2019-12-03; First posted 2019-12-06 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Upper Limb Surgery; Hand Surgery
Keywords: Articaine; Bupivacaine; Ultrasound; Supraclavicular block
MeSH Terms: interventions — Carticaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Articaine group (Experimental): Patients in this group are assigned to recieve 30 ml of Articaine 2%
  Interventions: Drug: Articaine
- Bupivacaine (Experimental): Patients in this group are assigned to recieve 30 ml of bupivacaine 0.5%
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Articaine — Supraclavicular block with 30 ml articaine 2%
  Other Names: Artinebsa
  Arms: Articaine group
Drug: Bupivacaine — Supraclavicular block with 30 ml bupivacaine 0.5%
  Other Names: Marcaine
  Arms: Bupivacaine

SUMMARY:
Effect of 2%Articaine versus 5%bupivacaine in pt undergoing short duration surgery in upper limb

DETAILED DESCRIPTION:
The investigator aim to compare Articaine 2% versus bupivacaine 0.5% in patient undergoing upper limb procedure under ultrasound guided supraclavicular block as regard onset and duration of sensory and motor block

ELIGIBILITY:
Inclusion Criteria:

* upper limb surgery
* ganglion removal
* k wiring
* Carapal tunnel

Exclusion Criteria:

* Coagulopathy.
* infection at site of injection.
* patient refusal.
* hypersensitivity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-03-22 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Duration of sensory block | Measured in minutes over 24 hours
  By pinprick test from 0 to 2 where 0 no sensory block and 2 complete anesthesia
Durations of motor block | Measured in minutes over 24 hours
  By Bromage scale from 1 to 4 where 1 no motor power and 4 full motor power
Duration of analgesia | Measured in minutes over 24 hours
  Measured by numerical analog scale where 0 no pain and 10 means worst pain

SECONDARY OUTCOMES:
Analgesia | 24 hours
  First analgesia required

CONTACTS AND LOCATIONS:
Overall Officials: Galal Mo El kadi, Doctor, Study Director — Professor
Locations (1):
- Ain Shams University hosptal, Cairo, Abbasya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data including primary and secondary outcome for all the participants
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 6 month after end of study
Access Criteria: Upon request from Corresponding Author

REFERENCES:
- [Derived] Armanious SH, Abdelhameed GA. A Randomized Controlled Trial: Comparison of 4% Articaine versus 0.5% Bupivacaine for Ambulatory Orthopedic Surgery under Supraclavicular Block. Anesthesiol Res Pract. 2020 Sep 24;2020:2194873. doi: 10.1155/2020/2194873. eCollection 2020. PMID 33029135